CLINICAL TRIAL: NCT00910351
Title: A Study to Evaluate the Safety and Pharmacokinetics of Ciprofloxacin in Adults and Children Aged 6 - 12 Years With Cystic Fibrosis Following Inhalation of Ciprofloxacin Dry Powder
Brief Title: Cipro Inhaler for Cystic Fibrosis Children Ages 6-12
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12759
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Pseudomonas Infection
Keywords: Cystic Fibrosis; Pharmacokinetics; Pediatrics; Inhalation; Sputum
MeSH Terms: conditions — Pseudomonas Infections; Cystic Fibrosis; Respiratory Aspiration | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro, BAYQ3939)

INTERVENTIONS:
Drug: Ciprofloxacin (Cipro, BAYQ3939) — 25 mg inhaled Ciprofloxacin

SUMMARY:
Ciprofloxacin PulmoSphere Inhalation Powder appears to be an effective and adequate antibiotic treatment for cystic fibrosis patients with P. aeruginosa colonisation. This planned study is the first study on the use of this new Ciprofloxacin PulmoSphere Inhalation Powder in the pediatric population of 6 to 12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with cystic fibrosis confirmed by genetic testing and / or by sweat test
* Colonization with P. aeruginosa confirmed in sputum in the past 12 months
* Cohort 1: greater than or equal to 18 years of age.
* Cohort 2: 6 - 12 years of age (inclusive)
* Normal Body Mass Index: BMI between 14.5 and 30 kg/m2, but in no case lower than the 30th percentile for age. Because CF patients are typically smaller than non-CF-patients, the normal body mass index will be based on standard CF foundation normal values for weight and sex.
* Patients who are able to understand and follow instructions and who are able to participate in the study for the entire period.
* Patients and legal representatives must have given their written informed consent to participate in the study after receiving adequate previous information and prior to any study specific procedures

Exclusion Criteria:

* Patients with FEV1 < 35% of predicted. FEV1 (forced expiratory volume) is a measure of lung function. This exclusion will prohibit enrollment of patients with severely impaired lung function.
* Patients with Burkholderia cepacia colonization of their respiratory tract
* Patients with acute bronchopulmonary aspergillosis (ABPA)
* Patients on a lung transplant list
* Patients with acute pulmonary exacerbations
* Patients with severe liver cirrhosis
* Massive hemoptysis in the preceding 4 weeks
* A history of relevant diseases of vital organs, of the central nervous system, or other organs not related to the underlying disease
* Patients with a history of severe allergies, non-allergic drug reactions, or multiple drug allergies
* Patients with hypersensitivity to the investigational drug or to other quinolones and/ or to inactive constituents
* Patients with known intolerance to hypertonic saline or bronchodilators
* Concomitant inhalation therapy with antibiotics and / or concomitant systemic therapy with fluoroquinolones
* Women who are pregnant

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of inhaled ciprofloxacin given as single inhalation dose to pediatric CF patients, aged 6 - 12 years | Two weeks post screening

SECONDARY OUTCOMES:
To investigate the pharmacokinetics of ciprofloxacin in plasma and sputum after inhalation administration | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (4):
  - Atlanta, Georgia
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Syracuse, New York